CLINICAL TRIAL: NCT05687097
Title: Untreated Sleep-related Breathing Disorders as an Aggravating Factor for Neuropathic Pain, Spasticity and Cardiovascular Dysfunction After Spinal Cord Injury: A Cross-sectional Prospective Study
Brief Title: Untreated Sleep Apnea as an Aggravating Factor for Other Secondary Medical Conditions After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Western University (Other)
Responsible Party: Principal Investigator, Julio Furlan, MD, Clinical Investigator and Scientist, University Health Network, Toronto
Other Study IDs: 19-5285
Record Dates: First submitted 2022-12-25; First posted 2023-01-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sleep Apnea; Spinal Cord Injuries; Spasticity, Muscle; Neuropathic Pain; Cardiovascular Complication
MeSH Terms: conditions — Sleep Apnea Syndromes; Spinal Cord Injuries; Muscle Spasticity; Neuralgia | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Individuals without sleep apnea after spinal cord injury: No significant sleep apnea is defined as an apnea-hypopnea index (AHI) < 5 events per hour of sleep
  Interventions: Device: Home-based sleep screening test or hospital-unattended sleep screening test; Device: Cardiovascular beat-to-beat monitoring; Device: ECG monitoring
- Individuals with mild sleep apnea after spinal cord injury: Mild sleep apnea is defined as an apnea-hypopnea index (AHI) ≥ 5 events per hour of sleep, but an AHI <15 events.
  Interventions: Device: Home-based sleep screening test or hospital-unattended sleep screening test; Device: Cardiovascular beat-to-beat monitoring; Device: ECG monitoring
- Individuals with moderate sleep apnea after spinal cord injury: Mild sleep apnea is defined as an apnea-hypopnea index (AHI) ≥ 5 events per hour of sleep but an AHI <15 events.
  Interventions: Device: Home-based sleep screening test or hospital-unattended sleep screening test; Device: Cardiovascular beat-to-beat monitoring; Device: ECG monitoring
- Individuals with severe sleep apnea after spinal cord injury: Severe sleep apnea is defined as an apnea-hypopnea index (AHI) > 30 events per hour of sleep.
  Interventions: Device: Home-based sleep screening test or hospital-unattended sleep screening test; Device: Cardiovascular beat-to-beat monitoring; Device: ECG monitoring

INTERVENTIONS:
Device: Home-based sleep screening test or hospital-unattended sleep screening test — ApneaLink device will be used to assess the number of apnea and hypopnea events per hour of sleep.
  Other Names: ApneaLink
Device: Cardiovascular beat-to-beat monitoring — CareTaker device will be used to continuously record the participant's arterial blood pressure and heart rate during sleep.
  Other Names: CareTaker
Device: ECG monitoring — Faror Bithium 180 device will be used to continuously record the participant's ECG during sleep.
  Other Names: Faros Bithium 180

SUMMARY:
This cross-sectional prospective study will assess the potential association of more severe sleep apnea after spinal cord injury with more intense neuropathic pain, more severe spasticity, and more significant cardiovascular abnormalities including cardiac arrhythmias and blood pressure fluctuations. In addition, the participants' experience when undergoing home-based sleep screening test or hospital-unattended sleep screening test will be assessed in a semi-structured interview.

DETAILED DESCRIPTION:
This cross-sectional prospective study will assess the potential association of more severe sleep apnea after spinal cord injury with more intense neuropathic pain, more severe spasticity, and more significant cardiovascular abnormalities including cardiac arrhythmias and blood pressure fluctuations. In addition, the participants' experience when undergoing home-based sleep screening test or hospital-unattended sleep screening test will be assessed in a semi-structured interview (qualitative analysis).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with subacute/chronic (> 1 month after injury) spinal cord injury.
* Individuals with a mid-cervical/mid-thoracic (levels C5 to T6) spinal cord injury.
* Individuals with a complete or incomplete (ASIA Impairment Scale A, B, C, or D) spinal cord injury.

Exclusion Criteria:

* individuals with other disorders of the central nervous system (e.g., sequelae of traumatic brain injury, stroke);
* Individuals with psychiatric disorders that can interfere with adherence to study;
* Individuals with neuromuscular diseases;
* Individuals with history of substance abuse;
* Individuals with prior history of hypersomnias or sleep apnea under treatment;
* Individuals with prior history of chronic pain (e.g. fibromyalgia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adults with subacute/chronic, cervical/thoracic, complete/incomplete SCI who were were not previously diagnosed with sleep apnea and under continuous positive airway pressure (CPAP) therapy at the time of the study enrollment and interventions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | One night of sleep (up to 10 hours)
  The number of apneas and hypopneas per hour of sleep recorded using the ApneaLink device.

SECONDARY OUTCOMES:
Neuropathic pain | Pre-intervention assessment only.
  Level of neuropathic pain prior to the interventions using Visual Analog Scale (0: no pain; 100: the worst pain ever).
Spasticity | Pre-intervention assessment only.
  Degree of spasticity prior to the interventions using the modified Ashworth Scale (0: normal tone; 16: all four extremities rigid in flexion or extension).
Cardiovascular dysfunction | Pre-intervention assessment only.
  The number of episodes of autonomic dysreflexia during sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Furlan, MD, Principal Investigator — KITE Research Institute, University Health Network
Locations (1):
- Lyndhurst Centre, TRI and KITE Research Institute, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared with another researcher when UHN REB approval is obtained.

REFERENCES:
- [Derived] Furlan JC, Loh E, Boulos MI. The potential effects of untreated sleep-related breathing disorders on neuropathic pain, spasticity, and cardiovascular dysfunction following spinal cord injury: A cross-sectional prospective study protocol. PLoS One. 2023 May 2;18(5):e0282860. doi: 10.1371/journal.pone.0282860. eCollection 2023. PMID 37130111